CLINICAL TRIAL: NCT00448851
Title: Phase 1 Study of Dermatophagoides Farinae Inhalation in Humans
Brief Title: Study of Dust Mite Inhalation in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David B. Peden, MD, Professor of Pediatrics, Director of CEMALB, University of North Carolina, Chapel Hill
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 06-0528; NHLBI-RO1 HL080337 (Other Grant/Funding Number: National Heart, Lung, and Blood Institute (NHLBI))
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Mild Asthma; Allergy
Keywords: asthma; allergy
MeSH Terms: conditions — Hypersensitivity; Asthma | interventions — Antigens, Dermatophagoides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): inhaled allergen challenge
  Interventions: Biological: inhaled allergen challenge

INTERVENTIONS:
Biological: inhaled allergen challenge — Subjects will inhale gradually increasing concentrations of Dermatophagoides farinae until a 15% drop in FEV1 is noted
  Other Names: dust mites

SUMMARY:
The purpose of this research study is to learn more about the effect of inhaled dust mite allergen extract on airway responses in allergic individuals with mild asthma. Information learned from this study will be used to identify a safe dose range of D Farinae extract for use in inhalation challenge studies. This study will also help determine how inhalation of the allergen affects mucociliary clearance (MCC) which is a measure of how quickly mucus clears from the airway.

DETAILED DESCRIPTION:
This will be a non-blinded study of the effect of inhaled house dust mite (D Farinae) allergen extract on airway responses, with the principal endpoint being a decrease in FEV1 of 15% within 10 minutes after inhalation of one of a sequence of doses of allergen compared with measurements obtained immediately prior to challenge. These doses will be delivered as 5 inhalations of allergen at concentrations of 0.25, 0.50, 1.0, 2.0, 4.0, 8.0, 16, 32, 64, 125, 250, 500, 1000, and 2000 AU/mL. Allergen challenge often induces an immediate and late phase decrease in lung function. The immediate phase that occurs within 10 minutes, often self resolves and is associated with release of histamine from airway mast cells, while the late phase response often occurs 2 to 8 hours later and is associated with increased airway inflammation.

During the subject's baseline visit occurring at least 2 days prior to allergen challenge, we will measure mucociliary clearance (MCC) of inhaled, radiolabeled particles by gamma scintigraphy. The subject will return 24 hours later for a follow-up scan and a sputum sample will also be collected. At 4 hours post allergen challenge, we will again measure MCC as an exploratory endpoint. It is expected that mucociliary clearance will be depressed as part of a late phase reaction to allergen challenge. Twenty-four hours after allergen challenge, induced sputum will be obtained and compared with the sputum sample obtained at the baseline visit. Exploratory endpoints of interest from examination of induced sputum will also be collected after inhaled allergen challenge.

Observation Schedule (details regarding study procedures follow below):

Baseline visit

1. Consent will be obtained
2. Review of subject's medical history and current medications
3. Vital sign measurements (temperature, pulse, respiratory rate, blood pressure), oxygen saturation, and symptom scoring
4. Urine pregnancy test for women of child bearing potential
5. Spirometry
6. Physical exam of the ears, nose, throat and chest
7. Xenon equilibrium gas scan
8. Mucociliary clearance procedure (MCC)

24 hours post baseline visit

1. Review any change in medical status over prior 24 hours
2. Vital signs, oxygen saturation and symptom score
3. Follow up MCC scan
4. Sputum induction

Post Challenge Observations/Reporting Subjects will be contacted for phone call follow-up 24 hours after sputum induction (see accompanying phone script)

24-48 hours prior to challenge visit (at least 2 days after the baseline visit)

1. Review any change in medical status since last visit
2. Vital signs, oxygen saturation, and symptom score
3. Spirometry
4. Physical exam of the ears, nose, throat and chest

Allergen challenge day

1. Review any change in medical status since last visit
2. Vital signs, oxygen saturation, and symptom score
3. Urine pregnancy test
4. Spirometry
5. If above measures are acceptable, allergen challenge will be performed as described
6. Post-challenge monitoring at intervals indicated on study worksheets
7. Four hours post challenge, subject will have MCC evaluated
8. Overnight stay in the UNC General Clinical Research Center (GCRC) Subjects will be instructed to perform either spirometry with a personal spirometer or peak flow assessments on an every other hourly basis until at least 9 pm, and up to 11 pm if the subject is awake.

24 hours post challenge

1. Subject is discharged from GCRC, and accompanied by a study staff member, proceeds directly to CEMALB.
2. Vital signs, oxygen saturation, and symptom score
3. Spirometry
4. Follow-up MCC scan
5. Sputum induction

Post Challenge Observations/Reporting

1. Subjects will be contacted for phone call follow-up 24 hours after post-challenge sputum induction (see accompanying phone script)
2. Each volunteer will be given a symptom scoring sheet for each day up to 96 hours (4 days) after challenge (see accompanying symptom scoring sheet)

Study discontinuation visit within 10 days of the final challenge dose:

1. Vital signs, oxygen saturation, and symptom score
2. Spirometry
3. If any findings are abnormal, medical evaluation as directed by the study physician will be undertaken

ELIGIBILITY:
Inclusion Criteria:

1. A history of episodic wheezing, chest tightness, or shortness of breath consistent with asthma, or physician diagnosed asthma.
2. Specific allergy to house dust mite Dermatophagoides farinae confirmed by positive immediate skin test response.
3. Provocative concentration of methacholine of 10 mg/ml or less producing a 20% fall in FEV1 (PC20 methacholine) by the method used in a separate screening protocol (98-CEMLB-293) that is already approved by the UNC IRB.
4. FEV1 of at least 80% of predicted and FEV1/FVC ratio of at least .70 (without use of bronchodilating medications for 12 hours), consistent with lung function of persons with mild episodic or mild persistent asthma.

Exclusion Criteria:

1. Any chronic medical condition considered by the PI as a contraindication to the exposure study including significant cardiovascular disease, diabetes requiring medication, chronic renal disease, or chronic thyroid disease.
2. Subjects with a history of immunologic disease, or undergoing therapeutic immune suppression for cancer or other diseases.
3. Physician directed emergency treatment for an asthma exacerbation within the preceding 12 months.
4. Use of systemic steroid therapy within the preceding 12 months for asthma or the following asthma symptoms; cough, wheeze, shortness of breath.
5. Use of inhaled steroids, cromolyn or leukotriene inhibitors (Montelukast or Zafirlukast) within the past month (except for use of cromolyn exclusively prior to exercise).
6. Use of daily theophylline within the past month.
7. Use of medications that might alter the response to methacholine or antigen challenge including anti-inflammatory and anti-histamine agents within one week of challenge.
8. Subjects using tricyclic antidepressants such as doxepin and MAO inhibitors.
9. Subjects using beta-adrenergic blockers or any other medications known to interfere with the treatment of anaphylaxis.
10. Inability to withhold inhaled or oral bronchodilating medications for 12 hours prior to allergen challenge.
11. Pregnancy (positive urine pregnancy test at the baseline visit) or nursing a baby. Pregnant women are excluded due to the risk of fetal exposure to radiation.
12. Women of child bearing potential who are not using dependable contraception (such as birth control pill, IUD, estrogen patches) or who are not completely abstinent.
13. Cigarette smoking >0.5 packs per week within the past 12 months.
14. Nighttime symptoms of cough or wheeze greater than 1x/week at baseline (not during a clearly recognized viral induced asthma exacerbation) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
15. Exacerbation of asthma more than 2x/week which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
16. Daily requirement for albuterol due to asthma symptoms (cough, wheeze, chest tightness) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma. (Not to include prophylactic use of albuterol prior to exercise).
17. Viral upper respiratory tract infection within 4 weeks of challenge.
18. Any acute infection requiring antibiotics within 2 weeks of challenge (or 4 weeks in the case of azithromycin due to the prolonged half-life).
19. Participating in any study utilizing an investigational agent within 4 weeks of this challenge.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2007-02; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Effect of allergen challenge procedure on the following:changes in airway monocytes cell surface marker expression and changes in airway PMN and Eosinophil numbers | 0-24 hours post challenge

SECONDARY OUTCOMES:
changes in symptom scores | day 0 through day 4 post challenge
changes lung function | 0-24 hours post challenge

CONTACTS AND LOCATIONS:
Overall Officials: David B Peden, MD, MS, Principal Investigator — University of North Carolina at Chapel Hill, Dept of Pediatrics / Center for Environmental Medicine, Asthma and Lung Biology
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Bennett WD, Herbst M, Alexis NE, Zeman KL, Wu J, Hernandez ML, Peden DB. Effect of inhaled dust mite allergen on regional particle deposition and mucociliary clearance in allergic asthmatics. Clin Exp Allergy. 2011 Dec;41(12):1719-28. doi: 10.1111/j.1365-2222.2011.03814.x. Epub 2011 Jul 5. PMID 21729182